CLINICAL TRIAL: NCT03190746
Title: Relationship of YWHAH Polymorphisms to Rheumatoid Arthritis Disease Severity
Status: Completed | Type: Observational
Sponsor: Keesler Air Force Base Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FKE 20150004H
Record Dates: First submitted 2017-06-11; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No SNP: Subjects have two copies of the wild type gene
  Interventions: Diagnostic Test: TaqMan SNP analysis
- SNP present: Subjects have one or two copies of the SNP
  Interventions: Diagnostic Test: TaqMan SNP analysis

INTERVENTIONS:
Diagnostic Test: TaqMan SNP analysis — TaqMan SNP analysis of the YWHAH gene

SUMMARY:
It is hypothesized that one or several of these 6 single nucleotide polymorphisms (SNPs) (rs2246704, rs2853884, rs3747158, rs4820059, rs7291050, and rs933226) in the YWHAH gene could be related to RA disease severity.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic inflammatory arthritis of substantial morbidity. Serum biomarkers such as Rheumatoid Factor and anti-cyclic citrullinated peptide assist with disease diagnosis and prognostic assessment of future disease activity. 14-3-3 eta is a relatively new RA serum biomarker. The 14-3-3 family of proteins were named based on chromatographic elution properites and are ubiquitously expressed intracellular chaperon proteins. The isoform relevant in RA is 14-3-3 eta. 14-3-3 eta provides additional information about RA to the clinician-it assists in making diagnosis, provides prognostic assessment of disease severity, and provides insight regarding response to therapy. Thus, 14-3-3 eta serves as an important mechanistic biomarker informing the clinician about patient's RA.

14-3-3 eta is the product of the YWHAH gene, located on chromosome 22q12.3. It is about 13 kilobase long, consisting of two exons separated by a single intron. This gene has been implicated in linkage studies to bipolar disorder and schizophrenia. Six YWHAH single nucleotide polymorphisms (SNPs) were identified in a prior study: rs2246704, rs2853884, rs3747158, rs4820059, rs7291050, and rs933226. rs2246704 was associated with bipolar disorder (Odds Ratio (OR) 1.31, p=0.03) and psychotic BP (OR 1.66, p=0.002). All six SNPs are intronic. It was hypothesized that one or several of these 6 single nucleotide polymorphisms (SNPs) could be related to RA disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Have RA per 1987 or 2010 American College of Rheumatology Classification Criteria

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients at an academic medical center
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Relationship to RA disease severity | 2.5 years
  The primary endpoint was the relationship of the six YWHAH SNPs to RA disease severity as based on the presence (1 point) or absence (0 points) across several domains: (A) serologic status (positive anti-CCP = 1 point, for example), (b) erosive changes (presence of erosions = 1 point), and (c) extra-articular manifestations (presence = 1 point).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Shaak, PhD, Study Chair — Research Director

IPD SHARING:
Plan to Share IPD: No
Small pilot trial with limited data